CLINICAL TRIAL: NCT06287359
Title: What is the Day-to-day Experience of Parents/Carers of Children or Adolescents With Severe Motor Disabilities Suffering From Spinal Pain?
Brief Title: Experience of Parents/Carers of Children With Severe Motor Disabilities Suffering From Spinal Pain?
Acronym: Vé-Quo-Pa-H-R
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2024/MP-01
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents/carers: Parents or carers of children with severe motor disabilities complaining of spinal pain
  Interventions: Other: individual interviews

INTERVENTIONS:
Other: individual interviews — Qualitative research with individual interviews

SUMMARY:
Parents of disabled children suffer from back pain more frequently than the general population. At present, the literature does not identify any specific factors responsible for this suffering.

For patients suffering from chronic back pain, there are specific treatment programmes in the Physical Medicine and Rehabilitation Department, with a focus on pain management.

The investigators would like to develop specific programmes for parents/carers of children/adolescents with severe motor disabilities.

To achieve this, it is important to gain a better understanding of the factors that contribute to the onset of pain.

With this in mind, the investigators are conducting a qualitative study to gain a better understanding of the day-to-day lives of these parents.

ELIGIBILITY:
Inclusion Criteria:

* Parents or carers of children with severe motor disabilities complaining of spinal pain

Exclusion Criteria:

* Parent/carer refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents or carers of children with severe motor disabilities complaining of spinal pain
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Individual interviews | baseline
  To understand the lived experience of parents/carers during the daily care of their child by means of a phenomenological analysis of the interviews

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes